CLINICAL TRIAL: NCT03829761
Title: Cerebellar Repetitive Transcranial Magnetic Stimulation (rTMS) for Reduction of Negative Affect and Treatment of Alcohol Use Disorder
Brief Title: Cerebellar Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jon Houck, Associate Professor of Translational Neuroscience, The Mind Research Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14918; R21AA026573 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2019-02-04 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder
Keywords: rTMS
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cerebellar rTMS (Experimental): Cerebellar rTMS. 1Hz repetitive transcranial magnetic stimulation (rTMS) to cerebellar vermis.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Sham TMS (Sham Comparator): Sham TMS. Sham transcranial magnetic stimulation to cerebellar vermis.
  Interventions: Device: Sham transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Repetitive transcranial magnetic stimulation (rTMS). Participants will undergo 10 daily sessions (Mon-Fri) of 30 minutes of 1Hz stimulation, for a total of 1800 pulses delivered.
  Arms: Cerebellar rTMS
Device: Sham transcranial magnetic stimulation — Sham transcranial magnetic stimulation (TMS). Participants will undergo 10 daily sessions (Mon-Fri) of 30 minutes of sham stimulation. Sham stimulation will imitate the active rTMS but does not have active stimulation.
  Arms: Sham TMS

SUMMARY:
The objective of the current study is to investigate the effects of repetitive transcranial magnetic stimulation (rTMS) on self-reported negative affect, cerebellar brain activation and alcohol use outcomes in alcohol use disorder (AUD).

DETAILED DESCRIPTION:
To achieve study aims, 34 treatment seeking adults with AUD will be recruited from local intensive outpatient (IOP) treatment programs and randomized to treatment with either inhibitory 1Hz rTMS to cerebellar vermis given daily for 2 weeks (total of 10 sessions) or sham. Alcohol use outcomes, self-reported negative affect, and craving will be obtained at baseline, 1 day, 1 week and 6 weeks following rTMS termination. An fMRI scan during a Stroop task will be obtained at baseline and 1 day after the final rTMS session.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-65 meeting DSM-V criteria for moderate or severe AUD in the past year;
* Interested in cutting down or quitting drinking;
* Able to provide voluntary informed consent;
* Have at least 4 heavy drinking days (≥ 5 drinks per day for men, and ≥4 for women) in the past 60 days;
* Currently receiving treatment for alcohol use disorder.

Exclusion Criteria:

* Severe neurological conditions (TBI/stroke/history of a seizure/dementia and other significant cognitive illnesses);
* Other urgent medical problems, as determined by the study physician from the history and physical exam;
* Schizophrenia, schizoaffective disorder, bipolar I disorder
* Suicidal thoughts (intent or plan) in the last month;
* Current moderate or severe other SUD (except nicotine or marijuana) or other drug (except nicotine or marijuana) use in the past month;
* Active legal problems with the potential to result in incarceration;
* Pregnancy or lactation, or child bearing age and sexually active but not on birth control (barrier methods allowed);
* Current daily use of anti-craving medications, antidepressants (at doses considered therapeutic for depression), benzodiazepines, antipsychotics (at doses considered therapeutic for psychosis or mood stabilization), mood stabilizers (at doses considered therapeutic for mood stabilization);
* Have previously undergone rTMS (to assure the blind is effective);
* Personal or familial (in first degree relatives) history of epilepsy;
* Any contraindication for Magnetic Resonance Imaging (MRI) or TMS including metal shards or certain implants (pacemakers etc.) in the body.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Time to drinking relapse as measured by the Time Line Follow Back | 8 weeks
  Time to drinking relapse as measured by the Time Line Follow Back from baseline in days.
Change in percent days abstinent as measured by the Time Line Follow Back | 3 weeks
  Change in percent days abstinent as measured by the Time Line Follow Back from the 90 days prior to day 1 to day 14-21 (post-treatment).
Change in self reported negative affect as measured by the Promise anger, anxiety and depression scales | 2 weeks
  Change in self reported negative affect as measured by the Promise anger, anxiety and depression scale T scores from baseline to day 15 (post-treatment).
Change in cerebellar brain activation as indicated by percent signal change in the medial cerebellum during incongruent minus congruent trials during a multisensory Stroop task during fMRI | 2 weeks
  Change in cerebellar brain activation as indicated by percent signal change in the medial cerebellum during incongruent minus congruent trials during a multisensory Stroop task during fMRI from baseline to day 15 (post-treatment). This will be calculated using a mask derived from preliminary data from a sample of 33 individuals with AUD at a single timepoint. Activation in this brain region was correlated with depression, anxiety, and recent drinking. Manuscript describing this result is under review (Wilcox et al.), and another manuscript describes the task in question (Wilcox et al. 2014 Cognitive Control Network Function in Alcohol Use Disorder Before and During Treatment With Lorazepam. Subst Use Misuse.

CONTACTS AND LOCATIONS:
Overall Officials: Jon M Houck, PhD, Principal Investigator — The Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No